CLINICAL TRIAL: NCT03319147
Title: Effect of Leucine-enriched Essential Amino Acid on Integrated Muscle Protein Synthesis and Muscle Recovery After Resistance Exercise
Brief Title: Effect of Amino Acid on Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EAA
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: exercise; recovery; muscle; protein
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 4g of maltodextrin
  Interventions: Dietary Supplement: Placebo
- Active (Active Comparator): 4g of essential amino acids
  Interventions: Dietary Supplement: Active

INTERVENTIONS:
Dietary Supplement: Active — 4g of essential amino acids
  Arms: Active
Dietary Supplement: Placebo — 4g of maltdextrin
  Arms: Placebo

SUMMARY:
The primary objective is to determine the impact of essential amino acids on integrated muscle protein synthesis over 4 days after resistance exercise.

In addition, the secondary objective is to determine the effect of essential amino acids on satellite cell regulation and inflammatory responses during this prolonged recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male, recreationally-active participants
* Healthy will be defined as screened by the PAR-Q+ (The Physical Activity Readiness Questionnaire for everyone; Appendix. B). Active will be defined as being in the top 20% of age specific scores on iPAQ (the International Physical Activity Questionnaire; Appendix.C).
* Participants are required not to engage in lower limb RT (resistance training) for at least 6 months prior to the study.
* Participants will be 18-35 years old.
* Participants are willing to abide by the compliance rules of this study

Exclusion Criteria:

* Female
* Inability to adhere to any of the compliance rules judged by principle investigator or medical doctor
* Self-reported regular tobacco use
* Self-reported illicit drug use (e.g. growth hormone, testosterone, etc.)
* The individual who has allergy for milk

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 4 hours
  Skeletal muscle fractional synthesis rate (%/h) will be determined by oral pulse method using ring-[D5]phenylalanine

SECONDARY OUTCOMES:
exercise performance | 4 days
  Maximal strength (torque in n-M) of the knee extensors will be assessed by a maximal isometric voluntary contraction (MVC).
Muscle soreness | 4 days
  Corresponding subjective ratings of muscle soreness will be collected from participants using a visual analogue scale (mm)
Muscle damage | 4 days
  Muscle damage will be determined by histochemical analysis. muscle damage is defined as Z-band streaming.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada